CLINICAL TRIAL: NCT04686981
Title: Vascular Surgery Department of Beijing Tsinghua Chang Gung Hospital
Brief Title: Endovascular thromBectomy of Acute Mesentery Vessels Occlusion Hybrid With Emergent Laparoscopic Surgery
Acronym: BOWEL
Status: Completed | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Weiwei Wu, Department director, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: 20283-0-01
Record Dates: First submitted 2020-12-16; First posted 2020-12-29 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Mesenteric Artery Ischemia; Thromboembolism
Keywords: Acute mesenteric artery thrombosis; Hybrid operation; Mechanical thrombectomy
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mesenteric artery thromboembolism patients: If all the radiography, physical signs, and laboratory markers hint at intestinal necrosis, exploratory laparotomy followed by enterectomy and thrombectomy is the first choice. If none of them hint at intestinal necrosis, endovascular therapy is superior. Laparoscopic exploration followed by endovascular therapy was performed for other patients, after that the intestinal blood supply was evaluated again by laparoscopy.

SUMMARY:
Acute mesenteric artery thromboembolism(AMT) is one of the important causes of acute abdomen and intestinal necrosis. If the intestinal blood supply is not restore in time, the prognosis of the disease is often poor and even endangers the life of the patient. Through laparoscopic surgery combined with modern minimally invasive endovascular technology, the blood supply of patients' intestine is restored. Observe the perioperative vascular patency rate, all-cause mortality, and the probability of short bowel syndrome. Through the hybrid operating room, we want to seek a multidisciplinary collaborative treatment mode to improve the long-term survival rate of such patients with enough intestines and completely free from TPN, and improve the prognosis of these patients.

DETAILED DESCRIPTION:
This study is a clinical cohort study; consecutively registered 30 patients with acute intestinal ischemia caused by superior mesenteric artery thromboembolism.

If all the radiography, physical signs, and laboratory markers hint at intestinal necrosis, exploratory laparotomy followed by enterectomy and thrombectomy is the first choice. If none of them hint at intestinal necrosis, endovascular therapy is superior. Laparoscopic exploration followed by endovascular therapy was performed for other patients, after that the intestinal blood supply was evaluated again by laparoscopy.

The main endpoints are the survival rate of bowel function preserved at 30 days, and the secondary endpoints are 30-day mortality, in-hospital mortality, symptoms-free survival rate, and rate of transition to laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intestinal ischemia and acute abdomen pain caused by superior mesenteric artery thromboembolism

Exclusion Criteria:

* Those who have acute large-area myocardial infarction, large-area cerebral infarction, or have serious heart failure or sequelae of cerebral infarction within 1 month;
* Combined with portal hypertension, gastrointestinal hemorrhage, portal and mesenteric venous reflux obstruction diseases;
* Contrast agent allergy, severe renal insufficiency, and inability to perform intravascular surgery;
* Past medical history contains superior mesenteric artery thromboembolism.
* Patients diagnosed with intestinal necrosis and peritonitis before surgery based on physical signs and imaging studies who directly undergo laparotomy and incision for thrombectomy.
* Patients without intestinal necrosis or peritonitis based on physical signs and imaging studies, who are treated by endovascular intervention therapy directly.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients suffering from superior mesenteric artery thromboembolism
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
survival rate with preserved bowel function | within 30 days after operations
  Counting data

SECONDARY OUTCOMES:
the incidence of all-cause mortality | within 30 days after operations
  Counting data
vascular patency rate | 180 days after operations
  Counting data

CONTACTS AND LOCATIONS:
Overall Officials: sifan yang, Study Director — Beijing Tsinghua Chang Gung Hospital
Locations (1):
- Beijing Tsinghua Chang Gung Hosipital, Beijing, Beijing Municipality, China